CLINICAL TRIAL: NCT05168241
Title: The Effect of Singing or Playing Melodica on Disease Symptoms, Self-Efficacy Level and Exercise Capacity in Chronic Obstructive Pulmonary Patients
Brief Title: The Effect of Singing or Playing Melodica in COPD Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, ELİF OKUR, PhD, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EOKUR
Record Dates: First submitted 2021-11-26; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; health promotion; musical instrument; singing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Singing; Control Groups

STUDY DESIGN:
Intervention Model Description: Power analysis was used to calculate the sample size of the study. The power of the test was calculated with the G*Power 3.1 program. The effect size was calculated as 1.24 according to the study of Canga et al., which was a similar study that was taken as a reference during the calculation process (28). The sample consisted of a total of 30 patients, 15 of whom were control and 15 were song/melodica, determined by power analysis at 95% confidence interval, 5% significance level and 1.24 effect size (df=28; t=1.701).
Masking Description: While taking informed consent, the purpose and content of the study were explained to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.the song/melodica group (Experimental): 15 patients in the song/melodica group. Pre-tests were applied to the song/melodica group in the first interview, and training was given according to Pender's Health Promotion Model. In addition to the trainings, the experimental group was given a total of 40 minutes twice a day, a total of 2 sessions, melodica training for the melodica group, and song activity for the singing group. In addition, the song/melodica group was encouraged to work at home for at least 20 minutes every day by providing the necessary motivation for singing or playing the melodica. The patient was asked to record his practices by keeping a diary.
  Two follow-ups were made by phone every 15 days, and the final tests were done face-to-face after 15 days. It tooks 10 weeks in total.
  Interventions: Other: song/melodica group
- 2. the control group (Other): 15 patients in the control group. The control group was given pre-tests in the first interview, they were trained according to Pender's Health Promotion Model, they were followed up twice every 15 days by phone, and the post-tests were done face-to-face after 15 days, It tooks 10 weeks in total.
  Interventions: Other: control group

INTERVENTIONS:
Other: song/melodica group — The patients who were divided into groups according to their wishes to sing or play the melodica were given warm-up training before the song group (20 min. warm-up training including breathing exercises, 20 min. singing) and melodica group (20 min. breathing). warm-up training including exercises, playing melodica for 20 minutes) was given with the researcher under the leadership of an experienced music teacher.
  For two weeks, a total of 40 minutes of song/melodica training was given per week. The singing group was given an assignment to sing for at least 20 minutes a day and the melodica playing group to play the melodica for at least 20 minutes a day. The patients were asked to do their song/melodica homework for at least 20-30 minutes a day, and then they were told about the follow-up papers.
  Patients in the song/melody group were followed up by telephone twice a total of 15 days at the 5th and 7th weeks.
  Other Names: singing or playing melodica
  Arms: 1.the song/melodica group
Other: control group — In the first interview, the pre-tests were applied by the researcher with the face-to-face interview technique. Afterwards, nursing education was given through the training guide prepared according to Pender's health promotion model. The control group was followed up and counseled by phone, twice a day, twice a day, in the 5th and 7th weeks.
  Post-tests were applied at week 10 to evaluate the effectiveness of the interventions.
  Other Names: Education according to Pender's health promotion model
  Arms: 2. the control group

SUMMARY:
This study was conducted as a randomized controlled experimental study to determine the effect of singing or playing melodica activity applied to chronic obstructive pulmonary patients on symptoms, self-efficacy level, and exercise capacity of patients.

DETAILED DESCRIPTION:
The research was carried out in the chest diseases polyclinics of a hospital in Trabzon city center between September 2020 and August 2021 with 30 patients: 15 in the control group and 15 in the song/melodica group. Based on Pender's health promotion model, the control group received training and counseling for ten weeks, including face-toface training and telephone follow-up. According to Pender's health promotion model, patients in the song/melodica group were given face-to-face training once, singing/playing the melodica training twice, and counseling and follow-up over the phone twice, with 15- day intervals. The data were collected with a patient information form and scales examining disease symptoms, self-efficacy, and exercise capacity. To evaluate the data, ttest, Mann-Whitney U, ANOVA, Kruskal Wallis test were used for independent groups to evaluate changes over time, and paired two-sample t-test, Wilcoxon test, and ANOVA test were used in repetitive measurements for dependent groups.

.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Having been diagnosed with COPD by the physician based on the results of the pulmonary function test taken with spirometry according to the GOLD criteria, who are in the stable period of COPD,
* Applying to thoracic polyclinics,
* not bedridden,
* Does not have vision and hearing problems that do not interfere with communication,
* Patients who can complete the six-minute walk test,
* Willing to sing and/or play melodica
* Patients who agreed to participate in the study and who read and signed the informed consent form were included in the sample.

Exclusion Criteria:-

* Those who do not agree to participate in the research,
* with asthma,
* with a diagnosis of cancer,
* with a diagnosis of Covid-19,
* Having unstable angina or myocardial infarction in the last 1 month,
* Having a resting heart rate >120/min,
* Patients with a resting systolic blood pressure of >180 mmHg and a diastolic blood pressure of >100 mmHg (183) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Modifiye Medical Research Council (mMMC) Dyspnea scale | 10 weeks
  Dyspnea scores of the patients were recorded in the pre-test and post-test.The Medical Research Council Scale (mMRC) consists of five items based on various physical activities that cause dyspnea.
  On this scale, patients are asked to simply select the activity that produces the feeling of dyspnea. Scoring is between 0-4. Minimum, maximum, median and mean values were evaluated for each group and compared between groups.

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | 10 weeks
  The CAT scale, which rates the effects of chronic obstructive pulmonary disease on the patient and deterioration in health, consists of eight parameters that question "cough, sputum, chest symptoms, fatigue, and confidence in leaving home".
  The score that can be obtained from the scale is a minimum of 0 and a maximum of 40 points. CAT scores of the patients were recorded in the pre-test and post-test. Minimum, maximum, median and mean values were evaluated for each group and compared between groups.

OTHER OUTCOMES:
six minutes walking tests | 10 weeks
  The 6-minute walking distances of the patients were recorded in the pre-test and post-test. Minimum, maximum, median and mean values were evaluated for each group and compared between groups.
COPD Self-Efficacy Scale | 10 weeks
  COPD Self-Efficacy Scale scores were recorded in the pre-test and post-test. A minimum of 34 points and a maximum of 170 points can be obtained from the scale as a total score. Minimum, maximum, median and mean values were evaluated for each group and compared between groups.
Hospital Anxiety Depression (HAD) Scale | 10 weeks
  Hospital Anxiety Depression (HAD) Scale scores were recorded in the pre-test and post-test.The answers are evaluated in a four-point Likert format and are scored between zero and three. The lowest score that can be obtained from both subscales is 0, and the highest score is 21. Minimum, maximum, median and mean values were evaluated for each group and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elif OKUR, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to share my individual participant data with other participants because I haven't published my work yet.

REFERENCES:
- [Background] Canga B, Azoulay R, Raskin J, Loewy J. AIR: Advances in Respiration - Music therapy in the treatment of chronic pulmonary disease. Respir Med. 2015 Dec;109(12):1532-9. doi: 10.1016/j.rmed.2015.10.001. Epub 2015 Oct 19. PMID 26522499
- [Background] Jones PW, Adamek L, Nadeau G, Banik N. Comparisons of health status scores with MRC grades in COPD: implications for the GOLD 2011 classification. Eur Respir J. 2013 Sep;42(3):647-54. doi: 10.1183/09031936.00125612. Epub 2012 Dec 20. PMID 23258783
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Wigal JK, Creer TL, Kotses H. The COPD Self-Efficacy Scale. Chest. 1991 May;99(5):1193-6. doi: 10.1378/chest.99.5.1193. PMID 2019177